CLINICAL TRIAL: NCT06415864
Title: Oral Cladribine B-cell Study
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 262436
Record Dates: First submitted 2024-04-03; First posted 2024-05-16 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cladribine (Mavenclad, Merck Serono Ltd): In the summary of product characteristics the recommended cumulative dose is 3.5 mg/kg body weight over 2 years, taken as 1 treatment course of 1.75 mg/kg per year. Each treatment course consists of 2 treatment weeks, 1 at the beginning of the first month and 1 at the beginning of the second month of the respective treatment year. Each treatment week consists of 4 or 5 days on which a patient takes 10 mg or 20 mg (1 or 2 tablets) as a single daily dose, depending on body weight

SUMMARY:
To study the impact of cladribine on peripheral and intrathecal B-cell, plasma cells, T cells and Tregs

DETAILED DESCRIPTION:
Primary: To quantify the temporal changes of memory B cells (CD19+/CD27+/IgD-/+), plasmablasts (CD19-/CD138+/CD38+) and T cells (CD4/CD45RA-/+, CCR7-/+, CD8+/CD45RA-/+/CCR7-/+), Tregs (CD4/CD8)/CD25+/CD127-/Fox3 P+) in the peripheral venous blood of pwMS with RRMS over 96w of treatment with oral cladribine.

These will be compared to the populations of non-memory or class-switched B cells (immature/transitional B cells CD10+/CD38+/CD19+, immature regulatory B cells CD10+/CD38+/CD19+/CD24+/IL-10+, mature B cells CD10-/CD38+/CD19+).

Secondary:

1. To study the effects of oral cladribine on:

   1. CSF OCBs and free immunoglobulin kappa and lambda light chain levels (FLC).
   2. CSF markers of inflammation, in particular CXCL-13 and urine markers of inflammation (neopterin).
   3. CSF markers of neuroaxonal damage, in particular free neurofilament light chains.
   4. On the peripheral repertoire B-cells (immunoglobulin) and T-cells (T cell receptor) and plasma cells (soluble receptors).
2. To compare CSF OCB positivity and CSF light chain levels with a contemporary control group of alemtuzumab treated pwMS (historical data).

Tertiary:

1. To compare B and T cell repertoire with a contemporary control group of alemtuzumab treated pwMS (historical data).
2. To evaluate the effect of changes in the immune cell profile on clinical measures of disability, MRI activity and PROMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MS who are being treated with oral cladribine at Barts Health NHS Trust will be approached to participate in this study.
* Patients must be willing and able to undergo lumbar punctures
* Patients who are OCB positive in their CSF (previous diagnostic lumbar puncture)

Exclusion Criteria:

* Ineligible for oral cladribine under NHS England prescribing guidelines and those participating in MAGNIFY-MS study (cladribine tablets in active MS)
* Unsuitable to have a lumbar puncture, for example spinal deformity, tethered cord syndrome or the use of aspirin or anticoagulants, and those unable to comply with study requirements, including frequency of visits and lumbar punctures.
* Presence of comorbidities in which the administration of cladribine is contraindicated.
* Abnormal baseline investigations (WBC<3 x 10*9/l, lymphocytes <1.0 x 10*9/l, neutrophil count <1.5 x 10*9/l, platelet count <100 x 10*9, haemoglobin <110g/l, LFT>/3x upper limit of normal of site reference ranges, potassium <2.8mmol/l or >5.5mmol/l, sodium <125 mmol/l, creatinine >130 umol/l)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Relapsing-remitting MS
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cladribine (Mavenclad, Merck Serono Ltd): In the summary of product characteristics the recommended cumulative dose is 3.5 mg/kg body weight over 96 weeks, taken as 1 treatment course of 1.75 mg/kg per year. Each treatment course consists of 2 treatment weeks, 1 at the beginning of the first month and 1 at the beginning of the second month of the respective treatment year. Each treatment week consists of 4 or 5 days on which a patient takes 10 mg or 20 mg (1 or 2 tablets) as a single daily dose, depending on body weight
Period: Overall Study
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 3 male, 7 female
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Class-switched Memory B Cells From Baseline to Week 96 nh
Description: Percent change from baseline to Week 96 in class-switched memory B cells (CD19+/CD27+/IgD-) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: B-cell and T-cell subsets were quantified by flow cytometry at baseline and Week 96. Percent change was calculated as [(Week 96 - baseline) / baseline] × 100.
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | -62.8 [-99.98 to 160]

2. Secondary Outcome: Changes in CSF of κ Free Light Chain (KFLC) From Baseline to Week 48 and Week 96
Description: The CSF κ Free Light Chain (KFLC) Index and λ Free Light Chain (LFLC) Index were measured at baseline, Week 48, and Week 96. KFLC and LFLC concentrations in cerebrospinal fluid and serum were obtained using Optilite. The KFLC Index and LFLC Index were calculated as (CSF FLC / serum FLC) ÷ (CSF albumin / serum albumin). These indices provide quantitative measures of intrathecal free light chain synthesis. Values are continuous laboratory measurements and do not use a score or scale.
Time Frame: Baseline to week 96
Measure: Mean (Standard Deviation); unit: kFLCIndex
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
kFLCIndex
  KFLC Index at baseline | 164.5 (227.1)
  KFLC Index at week 48 | 71.3 (82.74)
  KFLC Index at Week 96 | 64.4 (67.34)

3. Secondary Outcome: Change in CSF Oligoclonal Band (OCB) Positivity From Baseline to Week 48 and Week 96
Description: CSF and matched serum samples were analysed for IgG oligoclonal bands using isoelectric focusing followed by immunoblotting. OCB positivity was defined as ≥1 IgG band present in CSF but absent in serum (CSF-restricted bands). Reported values include the number of OCB-positive and OCB-negative participants at each time point (baseline, Week 48, Week 96). Higher values indicate increased intrathecal IgG synthesis
Time Frame: Baseline to week 96
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
Participants
  Participants with decreased OCB bands (Baseline → Week 96) | 4
  Participants with unchanged OCB bands | 2
  Participants with increased OCB bands | 3
  Participants OCB-negative at all timepoints | 1

4. Secondary Outcome: Changes in CSF of λ Free Light Chain (LFLC) Index From Baseline to Week 48 and Week 96
Description: as for outcome 2
Time Frame: Baseline to week 96
Measure: Mean (Standard Deviation); unit: LFLCIndex
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
LFLCIndex
  LFLC Index at baseline | 31.94 (25.47)
  LFLC Index at week 48 | 29.48 (25.14)
  LFLC Index at Week 96 | 27.18 (25.86)

5. Secondary Outcome: Change in CSF CXCL-13 Levels From Baseline to Week 96
Description: CXCL-13 concentrations in cerebrospinal fluid (CSF) were measured at baseline, Week 48, and Week 96 using immunoassay methods. Values are continuous laboratory measurements and are reported numerically (mean and standard deviation). No scoring system or clinical scale applies.
Time Frame: Baseline to week 96
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
pg/ml
  CXCL-13 at baseline | 88.6 (68.4)
  CXCL-13 at 48 weeks | 39.4 (35.2)
  CXCL-13 at 96 weeks | 19.1 (11.7)

6. Secondary Outcome: Change in Urine Neopterin Levels From Baseline to Week 96
Description: Urine neopterin concentrations were measured at baseline, Week 48, and Week 96 using immunoassay methods. Values are continuous laboratory measurements and are reported numerically (mean and standard deviation). No scoring system or clinical scale applied
Time Frame: Baseline to week 96
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
pg/ml
  Neopterin at baseline | 224.64 (268.06)
  Neopterin at 48 weeks | 355.87 (566.27)
  Neopterin at 96 weeks | 136.99 (114.18)

7. Primary Outcome: Percent Change in Non Class-switched Memory B Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in non class-switched memory B cells (CD19+/CD27+/IgD+) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | -85.3 [-99.98 to 134.44]

8. Primary Outcome: Percent Change in Plasmablast From Baseline to Week 96
Description: Percent change from baseline to Week 96 in plasmablasts (CD19+/CD27+/CD38+) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | 117.2 [-87.3 to 2250]

9. Primary Outcome: Percent Change in Transitional B Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in transitional B cells (CD19+ IgD+ CD10+ CD27-) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | 858.6 [-86.05 to 2350]

10. Primary Outcome: Percent Change in Regulatory B Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in regulatory B cells (CD19+/CD24+/CD38+) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | 648.3 [-93.52 to 46650]

11. Primary Outcome: Percent Change in CD4+ Central Memory T Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in CD4+ central memory T cells (CD45RA- CCR7+) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | -55 [-94.64 to 226.88]

12. Primary Outcome: Percent Change in CD4+ Naive T Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in CD4+ naive T cells (CD45RA+ CCR7+) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | -47.1 [-99.74 to 1472.97]

13. Primary Outcome: Percent Change in CD4+ TEMRA Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in CD4+ TEMRA cells (CD45RA+ CCR7-) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | 30.4 [-96.95 to 1560]

14. Primary Outcome: Percent Change in CD4+ Effector Memory T Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in CD4+ effector memory T cells (CD45RA- CCR7-) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | 0.82 [-96.90 to 234.25]

15. Primary Outcome: Percent Change in CD8+ Central Memory T Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in CD8+ central memory T cells (CD45RA- CCR7+) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
Percentage change | 26 [-94.24 to 251.57]

16. Primary Outcome: Percent Change in CD8+ Naive T Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in CD8+ naive T cells (CD45RA+ CCR7+) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | -25 [-89.67 to 2050]

17. Primary Outcome: Percent Change in CD8+ TEMRA Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in CD8+ TEMRA cells (CD45RA+ CCR7-) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | 60.81 [-52.84 to 3006.25]

18. Primary Outcome: Percent Change in CD8+ TEM Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in CD8+ effector memory T cells (CD45RA- CCR7-) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | 4.56 [-95.53 to 726.48]

19. Primary Outcome: Percent Change in Regulatory T Cells From Baseline to Week 96
Description: Percent change from baseline to Week 96 in regulatory T cells (CD4+ CD25+ FOXP3+) in participants with RRMS treated with oral cladribine.
Time Frame: Baseline to week 96
Population: as for outcome 1
Measure: Median (Full Range); unit: % change
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
% change | 40.02 [-88.52 to 680]

20. Secondary Outcome: Change in CSF Neurofilament Light Chain (NfL) Levels From Baseline to Week 96
Description: CSF neurofilament light chain (NfL) concentrations were measured at baseline, Week 48, and Week 96 using immunoassay methods. NfL is reported as a continuous laboratory value. Results are presented as numerical measurements (mean and standard deviation). No clinical scoring system or scale applies
Time Frame: Baseline to 96 weeks
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
pg/ml
  NFL at baseline | 534.42 [316.3 to 1249]
  NFL at 48wks | 271.77 [190.2 to 368.1]
  NFL at 96 wks | 301.13 [178.2 to 469.8]

21. Secondary Outcome: Change in CSF Soluble CD138 Levels From Baseline to Week 96
Description: Soluble CD138 concentrations in cerebrospinal fluid (CSF) were measured at baseline, Week 48, and Week 96 using immunoassay methods. Values are continuous laboratory measurements and are reported numerically (mean and standard deviation). No clinical scoring system or scale applies.
Time Frame: Baseline to week 96
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
pg/ml
  sCD138 at baseline | 0.25 (0.28)
  sCD138 at week 48 | 0.14 (0.20)
  sCD138 at week 96 | 0.09 (0.09)

22. Secondary Outcome: Changes in CSF Cytokine and Chemokine Levels From Baseline to Week 96
Description: Cerebrospinal fluid (CSF) cytokines and chemokines were measured at baseline, Week 48, and Week 96 using immunoassays. Analytes included IFN-γ, IL-10, IL-12p70, IL-13, IL-1β, IL-2, IL-4, IL-5, IL-8, and TNF-α. Values are continuous laboratory measurements and are reported numerically (mean and standard deviation). No clinical scoring system or scale applies. Results for each analyte are presented in separate rows of the results table.
Time Frame: Baseline to week 96
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
Number analyzed (Participants) | 10
pg/ml
  CSF IFN-y at baseline | 1.08 (0.75)
  CSF IFN-Y at 48 wks | 0.99 (0.90)
  CSF IFN-Y at 96 wks | 1.00 (1.22)
  CSF IL-10 at baseline | 0.11 (0.11)
  CSF IL-10 at 48 wks | 0.13 (0.19)
  CSF IL-10 at 96 wks | 0.05 (0.04)
  CSF IL12p70 at baseline | 0.015 (0.03)
  CSF IL12p70 at 48 WKS | 0.01 (0.01)
  CSF IL12p70 at 96 WKS | 0.02 (0.03)
  CSF IL13 at baseline CSF IL13 CSF IL13 baseline | 0.23 (0.27)
  CSF IL13 at 48 wks | 0.22 (0.24)
  CSF IL13 at 96 wks | 0.31 (0.20)
  CSF IL-1b at baseline | 0.11 (0.05)
  CSF IL-1b at 48wks | 0.11 (0.05)
  CSF IL-1b at 96wks | 0.08 (0.04)
  CSF IL-2 at baseline | 0.02 (0.03)
  CSF IL-2 at 48 WKS | 0.02 (0.03)
  CSF IL-2 at 96 WKS | 0.02 (0.02)
  CSF IL-4 at baseline | 0.0 (0.0)
  CSF IL-4 at 48wks | 0.0 (0.0)
  CSF IL-4 at 96wks | 0.0 (0.0)
  CSF IL-5 at baseline | 0.18 (0.09)
  CSF IL-5 at 48wks | 0.25 (0.13)
  CSF IL-5 at 96wks | 0.21 (0.14)
  CSF IL-8 at baseline | 27.11 (13.05)
  CSF IL-8 at 48 wks | 29.65 (9.56)
  CSF IL-8 at 96 wks | 25.56 (12.74)
  CSF TNF-a at baseline | 0.05 (0.04)
  CSF TNF-a at 48 wks | 0.04 (0.05)
  CSF TNF-a at 96 wks | 0.06 (0.06)

ADVERSE EVENTS:
Time Frame: 96 weeks
Description: In this observational study, adverse events (AEs) and serious adverse events (SAEs) are not collected in the same manner as interventional studies. Observational studies do not involve interventions administered as part of the research, and therefore, the definitions and reporting requirements for AEs and SAEs are not directly applicable.
Arm/Group | Cladribine (Mavenclad, Merck Serono Ltd)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT06415864/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT06415864/ICF_001.pdf